CLINICAL TRIAL: NCT04522154
Title: Transcatheter Tricuspid Valve Interventions and Right Ventricular Function: Evaluation with Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Principal Investigator, Muhammed Gerçek, Principal Investigator, Heart and Diabetes Center North-Rhine Westfalia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HDZ-KA_017_MG
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-01

CONDITIONS: Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MR-TTE (Other): Patient receiving cardiac magnet resonance imaging and echocardiography
  Interventions: Diagnostic Test: Magnet resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnet resonance imaging — Patients will receive a cardiac magnet resonance tomography before and 3-month after the procedure

SUMMARY:
There is an urgent need for transcatheter tricuspid interventions, as pharmaceutical therapy becomes ineffective in advanced disease stages and surgery remains associated with high mortality rates. Despite the promising results, in some patients, although good procedural results were achieved, no clinical improvements were measured. Right ventricular dysfunction is suspected to be the cause of the failed therapeutic strategy. Therefore this study aims to analyze right ventricular function with magnet resonance imaging before and 3-months after the procedure in order to gain insight into the prevalence and dynamics of right ventricular dysfunction in severe tricuspid regurgitation and to identify possible predictors for treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe tricuspid regurgitation undergoing transcatheter tricuspid intervention.

Exclusion Criteria:

* Patient with Incompatibility with magnetic resonance imaging or echocardiography
* Another valve disorder that requires treatment
* Severe precapillary pulmonary hypertension
* Unstable angina or percutaneous coronary intervention within the last 30 days
* Previous pacemaker/defibrillator implantation with intracardiac leads
* Patients with cardiac cachexia or a life expectancy less then 12 months
* Allergies to the material used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
Influence of transcatheter tricuspid intervention on tricuspid annular plane systolic excursion resonance tomography and echocardiography | 3 month
  Changes on tricuspid annular plane systolic excursion in magnet resonance tomography and echocardiography after of transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on right ventricular basal diameter excursion in resonance tomography and echocardiography | 3 Month
  Changes on right ventricular basal diameter in resonance tomography and echocardiography after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on right ventricular stroke volume resonance tomography and echocardiography | 3 Month
  Changes on right ventricular stroke volume in resonance tomography and echocardiography after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on right ventricular ejection fraction resonance tomography and echocardiography | 3 Month
  Changes on right ventricular ejection fraction in resonance tomography and echocardiography after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on right ventricular global longitudinal strain resonance tomography and echocardiography | 3 Month
  Changes on right ventricular global longitudinal in resonance tomography and echocardiography after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on right ventricular fractional area change resonance tomography and echocardiography | 3 Month
  Changes on right ventricular fractional area change in resonance tomography and echocardiography after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on tricuspid regurgitant fraction resonance tomography and echocardiography | 3 Month
  Changes on tricuspid regurgitant fraction in resonance tomography and echocardiography after transcatheter tricuspid intervention

SECONDARY OUTCOMES:
Exercise Testing with 6 min walking test | 3 month
  Changes on walked distance after transcatheter tricuspid intervention
rehospitalization rate | 3 month
  Detection of rehospitalization rate after transcatheter tricuspid intervention
Stroke | 3 month
  Detection of stroke rate after transcatheter tricuspid intervention
Death due to cardiovascular complication | 3 month
  Detection of death rate due to cardiovascular complications after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on the cardiopulmonary exercise capacity | 3 month
  Changes on aerobic capacity and endurance using the cardiopulmonary exercise testing (vO2max in milliliter per minute per kilogram)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Gercek, Dr. med., Principal Investigator — Assistant physician
Locations (1):
- Herz- und Diabeteszentrum, NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No